CLINICAL TRIAL: NCT02958137
Title: Arthroscopic Resection Arthroplasty of Basal Joint Arthritis: Comparing Outcomes of Isolated Carpometacarpal to Pantrapezial Disease
Brief Title: Arthroscopic Resection Arthroplasty of Carpometacarpal and/or Pantrapezial Osteoarthritis
Acronym: ARA:BJA-OA
Status: Completed | Type: Observational
Sponsor: Orthopaedic Specialist, PC, Davenport, IA (Other)
Responsible Party: Principal Investigator, Tyson Cobb, MD, Director of Hand and Upper Extremity Surgery, Orthopaedic Specialist, PC, Davenport, IA
Other Study IDs: Osquadcities
Record Dates: First submitted 2016-10-27; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Thumb Osteoarthritis
MeSH Terms: interventions — Arthroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Isolated CMC: Arthroscopic Resection Arthroplasty of isolated CMC joint OA. Please note, this is standard practice of Dr. Cobb's for treatment of CMC and/or STT arthritis.
  Interventions: Procedure: Arthroscopic Resection Arthroplasty
- Pantrapezial: Arthroscopic Resection Arthroplasty of simultaneous ARA of both the CMC and the STT joints. Please note, this is standard practice of Dr. Cobb's for treatment of CMC and/or STT arthritis.
  Interventions: Procedure: Arthroscopic Resection Arthroplasty

INTERVENTIONS:
Procedure: Arthroscopic Resection Arthroplasty — Surgical removal of the arthritic joint(s) using a minimally invasive technique.
  Other Names: Arthroscopy

SUMMARY:
Compare outcomes of ARA for isolated CMC OA versus to simultaneous ARA of CMC plus STT

DETAILED DESCRIPTION:
The purposes of this study were to report 1) long-term outcomes on a large series of patients that underwent arthroscopic resection arthroplasty (ARA) for thumb basal joint arthritis (BJA) and 2) to compare outcomes of ARA for isolated carpometacarpal osteoarthritis versus those undergoing simultaneous ARA of CMC plus the scaphotrapeziotrapezoid joint for pantrapezial disease.

Please note, all patients treated by Dr. Cobb for CMC and/or STT OA received the same treatment regardless of whether or not they chose to participate in the study. Patients who chose to enroll in the study received the same treatment as those who did not only their data was analyzed. Data collection is the same for those who do not participate, only their data is not analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Primary cases of ARA for thumb BJA with isolated CMC ARA or simultaneous ARA of the CMC and STT joints.

Exclusion Criteria:

* Exclusions included 19 cases that received interposition materials that since have been shown to produce unfavorable postoperative inflammatory responses, (Orthadapt Bioimplant, Pegasus Biologics, Irvine, CA and Artimplant Artelon CMC-I Spacer, Small Bone Innovations, LLC, New York, NY), 6 cases that had prior CMC surgery, and 27 cases that underwent concomitant surgeries that would potentially effect outcome.

Ages: 35 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients presenting with basal joint arthritis who were scheduled to undergo arthroscopic resection arthroplasty of the CMC and/or STT joints.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Strength (pinch and grip) | Change from baseline to 2 year follow-up.

SECONDARY OUTCOMES:
Satisfaction with Perceived Surgical Outcome | Reported at 2 year postoperative follow-up
  (0-5; 0 = not at all satisfied, 5 = completely satisfied)
Pain | Change from baseline to 2 year follow-up
  numerical rating scale, (0-10; 0 = no pain, 10 = worst imaginable pain)

IPD SHARING:
Plan to Share IPD: No
All patient health information was protected and complied with data privacy legal requirements. Personally identifiable patient information was removed from the data set prior to data analysis.